CLINICAL TRIAL: NCT03467334
Title: Nutritional Intervention, Multicenter, Randomized, Blind, Parallel Groups Study to Assess the Effect of Consumption of Bifidobacterium Breve CECT7263 and Lactobacillus Fermentum CECT5716 on Infant Colic
Brief Title: Infant Colic Treatment With Probiotics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mónica Olivares Martín; PhD (Industry)
Collaborators: European Regional Development Fund (Other); Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Sponsor-Investigator, Mónica Olivares Martín; PhD, Head of the R & D Department, Biosearch S.A.
Organization: Biosearch S.A. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P040
Record Dates: First submitted 2018-02-08; First posted 2018-03-16 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Infant Colic
Keywords: Infant colic; Bifidobacterium breve; Lactobacillus fermentum
MeSH Terms: conditions — Colic | interventions — Simethicone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The control group is the usual treatment that is administered differently (oral drops, 4 times a day) to the 2 research treatments (powder, 1 time a day).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- B. breve (Experimental): Group that will receive B. breve CECT7263 one dose per day in a capsule to open and suspend the powder in infant milk or water.
  Interventions: Dietary Supplement: B. breve
- B. breve plus L. fermentum (Experimental): Group that will receive B. breve CECT7263 and L. fermentum CECT5716 in one dose per day in a capsule to open and suspend the powder in infant milk or water.
  Interventions: Dietary Supplement: B. breve plus L. fermentum
- Simethicone 20 mg (Active Comparator): Control group that will receive simethicone 4 times (10 drops) a day.
  Interventions: Drug: Simethicone 20 MG

INTERVENTIONS:
Dietary Supplement: B. breve — Bifidobacterium probiotic strain at 1E+08 cfu/day
  Arms: B. breve
Dietary Supplement: B. breve plus L. fermentum — Probiotic combination at 2E+08 cfu/day
  Arms: B. breve plus L. fermentum
Drug: Simethicone 20 MG — Standard treatment for infant colic
  Arms: Simethicone 20 mg

SUMMARY:
This study evaluates the efficacy of Bifidobacterium breve CECT7263 and the mixture B. breve CECT7263/Lactobacillus fermentum CECT5716 in the treatment of infant colic. Group 1 will receive B. breve CECT7263 (2x10E8 CFU/day) one dose per day, group 2 will receive B. breve CECT7263 (1x10E8 CFU/day) and L. fermentum CECT5716 (1x10E8 CFU/day) in one dose per day, group 3 (control group) will receive simethicone 20 mg 4 times a day.

DETAILED DESCRIPTION:
Infant colic affects between 3-40% depending on the different criteria used for diagnosis. Recent studies carried out in healthy infants have shown that the consumption of B. breve CECT7263 and L. fermentum CECT5716 during the first months of life are related to a lower risk to present episodes of crying characteristic of infantile colic.

The objective of the present study is to compare the effect of B. brevis and B. brevis\L mixture. fermentum with respect to simethicone.

It is a multicenter, controlled, randomized, blind, parallel-group, 4-weeks nutritional intervention study which will be conducted in 18 public and private hospitals and health centers from Spain.

ELIGIBILITY:
Inclusion Criteria:

* Infants from 3 to 12 weeks of age
* Born at least at week 34
* Birth weight equal to or greater than 2000 grams
* Fulfill the criteria of Rome III
* Informed consent signed by parents or guardians

Exclusion Criteria:

* Failure to thrive
* Antibiotic treatment less than 2 weeks before the study or during the study
* Take probiotics as a treatment, different from the one that could contain the powdered infant formula
* Abandon breastfeeding and switch to infant formula
* Failure to comply with the study protocol

Ages: 3 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 156 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Crying time | 4 weeks
  Crying time in minutes per day

SECONDARY OUTCOMES:
Responders to treatment on weeks 1, 2, 3 and 4 | 4 weeks
  Number of responders to the treatment in each group on weeks 1, 2, 3 and 4. It is understood that responders are those infants who have experienced a daily decrease in the duration of the crises cries 50% above baseline
Gut microbiota | 4 weeks
  Effect of the treatment on intestinal microbiota: the levels of Escherichia coli, Clostridium, Bacteroides, Lactobacillus and Bifidobacterium at the beginning and at the end of the study (weeks 0 and 4) will be analyzed by quantitative PCR.
Stool carbohydrates | 4 weeks
  Stool carbohydrate levels: lactose and other carbohydrate levels will be analyzed by chromatography (Triple Quad LC/MS) at the beginning and end of the study (weeks 0 and 4).

CONTACTS AND LOCATIONS:
Overall Officials: José Maldonado, MD, PhD, Principal Investigator — Specialist in Pediatrics of the Medical-Surgical UGC of Infancy of the University Hospital Complex of Granada (Spain)
Locations (1):
- Servicio Andaluz de Salud, Granada, Spain